CLINICAL TRIAL: NCT00247637
Title: The Genetics of Endophenotypes and Schizophrenia
Brief Title: The Genetic Basis of Inherited Neurologic Deficits in People With Schizophrenia
Status: Completed | Type: Observational
Sponsor: University of California, San Diego (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Dr. David Braff, Professor, University of California, San Diego
Other Study IDs: R01MH065571 (NIH); R01MH065571 (NIH); R01MH065707 (NIH); R01MH065578 (NIH); R01MH065588 (NIH); R01MH065554 (NIH); R01MH065562 (NIH); DNBBS 7G-GRR
Record Dates: First submitted 2005-10-31; First posted 2005-11-02 (Estimated); Last update posted 2013-07-03 (Estimated); Status verified 2013-07

CONDITIONS: Schizophrenia
Keywords: Mental Health; Psychosis; Genetics; Heredity
MeSH Terms: conditions — Schizophrenia; Psychological Well-Being; Psychotic Disorders

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Whole blood was sent to the Cell Repository at Rutgers toestablish cell lines.

SUMMARY:
This is a study of the genetic basis of brain dysfunction in people with schizophrenia.

DETAILED DESCRIPTION:
Schizophrenia is a disabling disorder that is associated with specific inheritable neurobiologic deficits. These deficits can cause problems with memory, visual attention, information processing, and other aspects of daily living. Understanding the genetic components of these deficits in people with schizophrenia and their unaffected family members may help uncover the neurobiological basis, risk factors, and heritability of the disease. In addition, the information may serve to create more effective treatments and possibly a cure for the disease. This study will serve to provide information about the genetic basis of known inherited neurobiological deficits in people with schizophrenia. In turn, this may guide further studies on the genetics of schizophrenia.

Participants will attend 2 study visits, each of which will last approximately 4 hours. The first will include blood tests and diagnostic interviews of participating families to evaluate the presence of schizophrenic symptoms. The second study visit will entail four neurocognitive and neurophysiological tests. Participants will first have a pre-pulse inhibition test, which uses electrodes to measure eye blinking. Electrodes will also be placed on participants' head, ears, and around their eyes to measure brain waves. Next, participants will undergo an oculomotor test, during which they will wear glasses fitted with sensors that record eye movement. Participants will then be asked to repeat a list of words, letters, and numbers read by a researcher. Last, participants will undergo a computerized performance test requiring them to watch the computer screen and click a mouse whenever they see a number between 0 and 9. Each study visit will take approximately 4 hours.

ELIGIBILITY:
Inclusion Criteria for Participating Families:

* Families with at least one member who has schizophrenia

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The subject population will include schizophrenia probands (12 per site per year), first degree relatives (36 per site per year) and normal comparison subjects (15 per site per year). The proband must meet the diagnosis of schizophrenia by DSM-IV criteria. There must be at least one parent and one unaffected sibling in the pedigree. Therefore a total of 315 subjects will be enrolled at each site each year with a total of 2205 enrolled across all 7 sites. Schizophrenia probands and normal subjects will be between 18 and 65 years of age. Exclusion criteria include visual or hearing impairments, history of head trauma, organic brain dysfunction, neurological disease, and significant drug or alcohol use and for controls, significant psychiatric history and/or current use of psychotropic medications. We will include equal numbers of men and women and all appropriate subjects willing to participate regardless of ethnic background.
Sampling Method: Non-Probability Sample
Enrollment: 2025 (Actual)
Dates: Start 2003-05; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
percent inhibition to the 60 msec prepulse, P50 suppression, proportion of correct saccades, d, number correct in the reorder condition, the total recall score | Upon entry to the study
  The primary outcome measure for each endophenotype is as follows: for prepulse inhibition (PPI) the primary measure is the percent inhibition to the 60 msec prepulse; for P50 suppression it is the difference in amplitude between the test and conditioning stimuli; for antisaccade it is the proportion of correct saccades; for the DS-CPT it is (d') which is based on correct target detections and incorrect responses to nontargets; for LNS it is the number correct in the reorder condition; for CVLT it is the total recall score summed across 5 trials.

CONTACTS AND LOCATIONS:
Overall Officials: David Braff, MD, Study Director — University of California, San Diego
Locations (7):
- United States (7):
  - University of California Los Angeles, Los Angeles, California
  - University of California, San Diego, San Diego, California
  - University of Colorado Health Sciences Center, Denver, Colorado
  - Harvard University, Boston, Massachusetts
  - Mount Sinai School of Medicine, New York, New York
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Washington and VA Puget Sound Health Care System, Seattle, Washington

REFERENCES:
- See also: Click here for more information on the Schizophrenia Research Program — http://www.schizophreniaresearch.net